CLINICAL TRIAL: NCT06501950
Title: Measuring Silent Disease Progression in Multiple Sclerosis With a Multimodal Approach
Acronym: 360PMS
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Dr. med. Marc Günter Pawlitzki, Study coordinator / PI, Heinrich-Heine University, Duesseldorf
Other Study IDs: 360PMS_1.0
Record Dates: First submitted 2024-06-20; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Follow-Up; Observational study; PIRA; RRMS; PPMS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Core centre: Persons that will be included by the core centre will be examined every 6 months by clinical testing, blood tests, and optical coherence tomography. A MRI will be conducted every 12 month. Additional digital monitoring using a smartwatch and smartphone ist optional.
- Other study centre: Persons that will be included by the other study centre will be examined every 6 months by clinical testing and blood tests. Additional digital monitoring using a smartwatch and smartphone ist optional.

SUMMARY:
This observational study wants to examine the disease progression independent of relapses in patients with Multiple Sclerosis (MS) that are treated with monoclonal antibodies. Participants will be clinically examined every 6 months and optionally receive a magnetic resonance imaging (MRI) every 12 months. The investigators will also take blood for blood biomarker tests with each clinical examination. Optionally, digital data can be continuously collected via smartphone and smartwatch.

With this information the study will compare the results from clinical, digital, radiological, and blood-based tests with the disease progression the participants report themselves. This study aims to investigate what percentage auf patients with MS under antibody treatment experience a slow progression of the disease.

DETAILED DESCRIPTION:
The goal of this observational prospective, observational, multicenter proof of concept study is to identify silent disease progression in people with multiple sclerosis (MS) that are treated with monoclonal antibodies.

Progression independent of relapse activity (PIRA) refers to disability progression unrelated to relapses. Treatment with disease-modifying agent shifts the primary cause of disability towards PIRA, likely due to the prevention of relapses during therapy. In order to promptly identify these patients in the future, newer biomarkers are needed that can detect disease activity more sensitively. Digital health technologies (DHTs), such as connected wearables, offer the capability of continuously collecting real-life data. As they can capture movement patterns, sleep behavior, and cognition, DHTs can document silent disease progression in MS patients and have the potential to enhance our understanding of disease activity.

The goal of the 360 PMS (progressive Multiple Sclerosis) study is to evaluate various widely available smartwatch-derived digital metrics and blood-based analyses as well as imaging tools for monitoring silent disease activity in MS patients at two study centres. Patients with relapsing remitting or primary progressive MS that are treated with monoclonal antibodies and do not have an Expanded Disability Status Scale (EDSS) of more than 7,0 will be included in this study.

Clinical evaluations will be conducted every 6 months, as well as blood-based measurements that include serum neurofilament-light-chain (sNfL), glial fibrillary acidic protein (GFAP) and proteomic data. Data captured by smartwatches (Withings Scanwatch) include activity-related data (step count, minutes in certain intensity levels), basic cardiovascular measurements such as heart rate, and sleep-related data (total time asleep, sleep efficiency and quality etc.). Additionally, disease progression can be optionally evaluated by monitoring fine motor skills while typing on the smartphone by a smartphone application (Neurokeys).

The study will initially start at the core centre at the University Clinic Düsseldorf and plans to enrol further sites in the months following initiation. Further centers might not include optical coherence tomography (OCT) or MRI measurements. At the core facility additional examinations will be conducted: Structural MRI examinations will be conducted at baseline and in month 12 and 24. OCT measurements will examine retinal morphology and be conducted every 6 months.

The investigators will attempt to closely analyze MS patients under treatment with monoclonal antibodies with these methods. Data will be collected for a 24-month prospective period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS or PPMS according to the 2017 McDonald criteria
* Current treatment with monoclonal antibodies (including Natalizumab, Ofatumumab, Ocrelizumab) according to SmPC
* EDSS ≤7.0

Exclusion Criteria:

* Patients with an acute MS relapse and/or a history of intravenous corticosteroid treatment within past six weeks.
* Any comorbidity resulting in an impairment to understand or successfully complete the study such as (but not restricted to) psychiatric comorbidities or dementia. Decision will be made at investigators discretion.
* Additional immunosuppression except of above mentioned monoclonal antibodies
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RRMS or PPMS that are currently treated with a monoclonal antibody.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Progression independent from relapse (PIRA )at month 24 | Baseline up to 24 months
  Composite confirmed disability accumulation (CDA) defined as disability increase from study baseline, measured by Expanded Disability Status Scale (EDSS) (an increase of ≥1.0 points if baseline EDSS was ≤5.5 points or an ≥0.5-point increase if baseline EDSS)was >5.5 points) or an increase of 20% of more in Timed 25-Foot Walk (T25FW) or an increase of 20% or more in Nine-Hole Peg Test (9HPT) confirmed at the subsequent study visit (minimum acceptable interval 12 weeks). Composite relapse-associated worsening (RAW) events are defined as a subset of composite CDA events. In these, the initial disability increase from study baseline occurred 90 or fewer days after the onset of a relapse

SECONDARY OUTCOMES:
EDSS: Change From Baseline in Expanded Disability Status Scale (EDSS) Score | Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The EDSS is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Higher scores indicate the worse level of disability.
Change From Baseline in World Health Organization Quality of Life Brief Version (WHOQOL-BREF) Score | Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The WHOQOL-BREF questionnaire measures quality of life across 4 domains: Physical health, psychological health, social relationships and environment. It also includes one question on overall QOL and one on general health. The WHOQOL-BREF scores correlate highly (.89 or above) with WHOQOL-100 scores, and demonstrate good discriminant validity, content validity, internal consistency and test-retest reliability. The four WHOQOL-BREF domain scores will be used as main outcome measure. The measure is calculated by summing the point values for the questions corresponding to each domain and then transforming the scores to a 0-100 point interval, higher score correspond to greater QOL.
Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score - Component Paced Auditory Serial Addition Test | Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The Paced Auditory Serial Addition Test (PASAT) measures cognitive processing speed and working memory by evaluating how accurately participants can perform mental arithmetic tasks while listening to a series of numbers. It's one of the components of the Multiple Sclerosis Functional Composite (MSFC), alongside the Timed 25-foot walk (T25FW) and the 9-hole peg test (9HPT) for both dominant and nondominant hands. The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes.
Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score - Component 9-hole peg test | Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The 9-hole peg test (9HPT) evaluates manual dexterity by assessing the time it takes for a participant to complete the task using both dominant and nondominant hands. It's part of the Multiple Sclerosis Functional Composite (MSFC), which also includes the Timed 25-foot walk (T25FW) and the Paced Auditory Serial Addition Test (PASAT). The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes
Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score - Component Timed 25-foot walk (T25FW) | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The Timed 25-foot walk (T25FW) assesses mobility and ambulation by measuring the time it takes for a participant to walk 25 feet. It's a component of the Multiple Sclerosis Functional Composite (MSFC), along with the 9-hole peg test (9HPT) for both dominant and nondominant hands, and the Paced Auditory Serial Addition Test (PASAT).
  The MSFC Z-score is calculated by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score. A Z-score represented the number of standard deviations participant's test result was higher (Z >0) or lower (Z <0) than the average test result (Z = 0) from the reference population. Higher scores indicate better outcomes
Change in Pittsburgh Sleep Quality Index (PSQI) | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality and disturbances over a one-month period. It comprises 19 items covering seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  The PSQI global score is calculated by summing the scores of these components, resulting in a range from 0 to 21. Higher scores indicate worse sleep quality, with scores ≥ 5 denoting poor sleep quality.
Change From Baseline in Fatigue Severity Scale (FSS) | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  The FSS is a self-assessment questionnaire that provides a score as a measurement of the severity of fatigue. It consists of 9 questions scored from 1 to 7, low value indicates strong disagreement with the statement, whereas a high value indicates strong agreement. A total score of 36 or more suggests the presence of fatigue.
Change in blood-based serum filament lightchain (sNFL) levels | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  As measured by Roche's Elecsys NfL kit in pg/ml from serum samples.
Change in blood-based glial fibrillary acidic protein(GFAP) levels | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  As measured by Roche's Elecsys NfL kit in pg/ml from serum samples.
Change in proteomic signatures | Time Frame: Baseline up to 24 months (after 6 months, 12 months, 18 months, 24 months)
  As determined by serum-based proteomics. Comparisons will focus on correlations between protein expression and other clinical and paraclinical markers.
Questionnaire about smartwatch usage (System Usability Score) | After 6 months and 24 months of use]
  The System Usability Scale (SUS) evaluates the usability of various systems, including software applications, websites, and user interfaces. It consists of a 10-item questionnaire with five response options ranging from Strongly Agree to Strongly Disagree.
  The SUS score is calculated by summing the item scores and converting them to a range from 0 to 100. Higher scores indicate better usability. The SUS provides a global view of subjective usability assessments, applicable to a wide range of design products and services, including healthcare systems and applications.
Changes in fine motor skills composite as calculated by Neurokeys | Through study completion, up to two years
  The smartphone application Neurokeys examines the users' skills while typing with its digital keyboard and collects data on the users longitudinal development of fine motor skills. Measurements are based on a proprietary algorithm that takes in account time of flight while typing and other measurements.
Changes in cognition composite as calculated by Neurokeys | Through study completion, up to two years
  The smartphone application Neurokeys examines the users' typing and information processing skills and subsequently calculates a cognition composite score using a proprietary algorithm.
Wearing time of smartwatch (daily) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch and the associated HealthMate smartphone application.
Longitudinal development of activity parameter: step count | Continuously during the entire observation period
  Measured by the smartwatch Withings Scanwatch and the associated HealthMate smartphone application.
Longitudinal development of activity parameter: approximate distance traveled (meter) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of activity parameter: duration of soft activity (seconds) defined by Withings | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of activity parameter: duration of moderate activity (seconds) defined by Withings | Continuously during the entire observation period (up to 24 months)
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of activity parameter: duration of intense activity (seconds) defined by Withings | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of activity parameter: sum of all active time (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: time awake (seconds) | Continuously during the entire observation period (24 months)
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of activity parameter: approximate calories burned | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: number of times user woke up | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: time to sleep (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: heart rate variability (ms) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: total time asleep (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: total time in bed (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: ratio of sleep/time in bed | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: time spent in bed before falling asleep (seconds | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: time awake after first falling asleep (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of sleep parameter: Withings Sleep score | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: maximal heartrate | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: minimum heartrate | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: time in light heartrate zone (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: time in moderate heartrate zone (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: time in intense heartrate zone (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2
Longitudinal development of cardiovascular parameter: time in maximal heartrate zone (seconds) | Through study completion, up to two years
  Measured by the smartwatch Withings Scanwatch 2

CONTACTS AND LOCATIONS:
Overall Officials: Marc Günter Pawlitzki, PD Dr. med., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Düsseldorf, Department of Neurology, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kappos L, Wolinsky JS, Giovannoni G, Arnold DL, Wang Q, Bernasconi C, Model F, Koendgen H, Manfrini M, Belachew S, Hauser SL. Contribution of Relapse-Independent Progression vs Relapse-Associated Worsening to Overall Confirmed Disability Accumulation in Typical Relapsing Multiple Sclerosis in a Pooled Analysis of 2 Randomized Clinical Trials. JAMA Neurol. 2020 Sep 1;77(9):1132-1140. doi: 10.1001/jamaneurol.2020.1568. PMID 32511687
- [Background] Masanneck L, Voth J, Huntemann N, Ozturk M, Schroeter CB, Ruck T, Meuth SG, Pawlitzki M. Introducing electronic monitoring of disease activity in patients with chronic inflammatory demyelinating polyneuropathy (EMDA CIDP): trial protocol of a proof of concept study. Neurol Res Pract. 2023 Aug 24;5(1):39. doi: 10.1186/s42466-023-00267-3. PMID 37612774